CLINICAL TRIAL: NCT03105687
Title: A Multicenter, Assessor-blinded, Controlled, Randomised, Parallel Group, Superiority, Pragmatic Trial Assessing the Effectiveness of Daily SMS-reminders in Pharmaceutical Care of Older Adults With Hypertension on Improving Patients' Adherence to Blood Pressure-lowering Medication
Brief Title: Effectiveness of SMS Reminders of Blood Pressure-lowering Drugs Intake
Acronym: SPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Collaborators: University of California, Los Angeles (Other); Research Institute for Child Psychology and Pathopsychology (Unknown); Dr. Max Pharmacies (Unknown)
Responsible Party: Principal Investigator, Zuzana Haramiova, PharmDr., Comenius University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SPPA-2017
Record Dates: First submitted 2017-03-17; First posted 2017-04-10 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Hypertension; Primary Hypertension; Non-Adherence, Medication; Non-Adherence, Patient
Keywords: mHealth; SMS reminders; adherence; antihypertensive drugs; pharmacists; cost-effectiveness
MeSH Terms: conditions — Hypertension; Essential Hypertension; Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the Control group will receive standard Pharmaceutical Care according to the principles of Good Pharmaceutical Practice and national Slovak legislation requirements only.
  Participants in the control group will also receive a welcome SMS one day after enrollment and an end-of-trial SMS three months after the enrollment. Additionally, prior to their scheduled follow-up visit (Visit 2), three months following the enrollment, trial pharmacists will call the participants to remind them of their follow-up visit.
- Intervention (Experimental): Participants in the intervention group will also receive standard Pharmaceutical Care provided by the trial pharmacist, the welcome SMS and the end-of-trial SMS. Additionally, they will receive daily SMS reminders of their blood pressure-lowering medication intake from a trial pharmacist for a period of 3 months after the enrollment. The structure of the SMS reminder will follow the information provided as a part of the usual drug dispensation and counselling process as described in the Slovak national Decree No. 129/2012 Coll. Thus, most of the data are available on the prescription and all of the collected data are already a well-established and required part of the standard Pharmaceutical Care in Slovakia. The simple structure of the SMS reminder will allow for future reproducibility.
  Interventions: Behavioral: SMS reminders of medicines intake

INTERVENTIONS:
Behavioral: SMS reminders of medicines intake — The intervention consists of daily SMS reminders of blood pressure-lowering medication provided by a pharmacist for a period of 3 months.
  Arms: Intervention

SUMMARY:
By conducting the SPPA trial we try to find out, whether personalized Short Message Service (SMS) reminders of blood pressure-lowering medication can effectively increase patients' adherence to blood pressure-lowering medication. Additionally, we also evaluate their effect on patients' systolic blood pressure control.

DETAILED DESCRIPTION:
Hypertension belongs to the main risk factors of cardiovascular diseases, which are the leading cause of morbidity and mortality in the world and in the Slovak Republic. Despite the availability of effective antihypertensive treatment, blood pressure control remains a serious problem. Poor adherence to blood pressure-lowering medication is considered to be the key factor for uncontrolled blood pressure. Studies estimate the overall adherence to medication in patients with chronic diseases at around 50%. Slovak studies report even significantly lower adherence rates (15-19%), which underlines the urgency to address this health problem in the Slovak Republic. The majority of interventions aimed at increasing patients' adherence are associated with substantial costs and health care professionals capacity, both lacking in the current Slovak health care system. Several studies have shown the efficiency of SMS reminders to improve patients' adherence and health outcomes at very low cost. Since mobile phones are frequently used among Slovak inhabitants and SMS messages are a popular mean of communication, this approach could be feasible also in Slovakia. Pharmacists are highly trained drug experts who have the knowledge, skills and time to address patients' nonadherence using a simple SMS reminder system.

Thus, our research question is as follows: Do personalized daily SMS reminders of blood pressure-lowering medication intake provided by pharmacists in addition to standard Pharmaceutical Care reduce the proportion of nonadherence to blood pressure-lowering medication among older ambulatory patients with hypertension in Slovakia? And we hypothesize that personalized daily SMS reminders of blood pressure-lowering medication intake provided by pharmacists in addition to standard Pharmaceutical Care increase the proportion of adherence to blood pressure-lowering medication among older ambulatory patients with hypertension in Slovakia from 30% to 49% in the intervention group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years (from the day of the 55. birthday inclusive)
* Diagnosis of primary (essential) hypertension (I10 according to International Classification of Diseases (ICD-10))
* Filling of blood pressure-lowering prescription(s) at trial recruitment (Visit 1)
* Duration of antihypertensive drug treatment for at least 1 year without any discontinuation
* Ownership of a mobile phone for personal use with the ability to open and read SMS
* Understanding of Slovak language on native-speaker level
* Informed consent for participation in the clinical trial and personally signed Informed Consent Form

Exclusion Criteria:

Exclusion criteria assessed prior to patient enrolment (by trial pharmacists):

* Planned hospitalisation during the trial period (3 months)
* Biological impairment affecting the ability to read the SMS (e.g. loss of vision, visual field cuts, aphasia)
* Living in the same household with another trial participant
* Participation in another clinical trial

Exclusion criteria assessed after patient enrolment (by trial pharmacists and project leader):

* Hospitalisation during the trial period
* Patient informs he/she won't be able to participate in the trial
* Withdrawal of Informed Consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Combined adherence endpoint | at Visit 2 (follow-up visit after 3 months of intervention period)
  Measurement variable: adherence status (dichotomous) assessed via the eight item Morisky Medication Score (MMAS-8) as follows:
  adherent: MMAS-8 score ≥6 and pill count rate ≥80% or <=120% non-adherent: MMAS-8 score <6 and/or pill count rate <80% or >120% Analysis Metric: final value (Visit 2) Method of aggregation: proportion of adherent patients (%)

SECONDARY OUTCOMES:
Change in medians of MMAS-8 after 3 months | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  Specific measurement variable: MMAS-8 (categorical, ordinal) Analysis Metric: change from baseline (Visit 1) Method of aggregation: median
Mean Adherence Rate (%) after 3 months calculated via pill count | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  Specific measurement variable: adherence rate (%), continuous variable Analysis Metric: final value (at Visit 2) Method of aggregation: mean
Mean change in systolic BP after 3 months | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  Specific measurement variable: systolic blood pressure in mmHg (continuous variable) Analysis Metric:change from baseline (Visit 1) Method of aggregation: mean
Patients' satisfaction with SMS reminders. | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  Patient satisfaction will be assessed using a Satisfaction Questionnaire based on previous studies.

OTHER OUTCOMES:
Overall direct treatment costs | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  Direct treatment costs (monthly average) of blood pressure-lowering medication for each patient will be assessed according to the List of categorized drugs issued by the Ministry of Health of the Slovak Republic.
Signals of adverse events associated with blood pressure-lowering medication | at Visit 2 (at follow-up visit; 3 months after Visit 1)
  During the whole course of the trial we will actively seek for signals of adverse events associated with blood pressure-lowering medication. Patients will have te possibility to report them any time during the trial. Additionally, trial pharmacists will specifically ask the patients about any potential signals of adverse events at Visit 2.
Number of patients who refused to participate in the study (Patients Refusal Rate) | Trough enrollment
  We will collect the number of patients who refused to participate in the study and report it as percentage of the overall approached patients.
Number of participants who withdrew from the study (Participants Withdrawal Rate) | From date of randomization until Visit 2 (3 months after Visit 1) or the date of early study termination, whichever came first, assessed up to 3 months
  We will collect the number of patients who withdrew from the study (early study termination) and report it as percentage of the overall study participants. Also, anonymous reasons for withdrawal from study will be collected, if the patients wish to provide such information.

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Haramiova, PharmDr., Study Director — Faculty of Pharmacy Comenius University in Bratislava, Department of Organization and Management of Pharmacy; Magdalena Kuzelova, Prof., PharmDr., PhD., Study Chair — Faculty of Pharmacy Comenius University in Bratislava, Department of Pharmacology and Toxicology; Donald M. Morisky, Sc.D., M.S.P.H., Sc.M., Study Chair — Fielding School of Public Health, Department of Community Health Sciences; Tomas Tesar, Doc., PharmDr., PhD, MBA, Study Chair — Faculty of Pharmacy Comenius University in Bratislava, Department of Organization and Management of Pharmacy; Michal Stasko, PharmDr., Study Chair — Faculty of Pharmacy Comenius University in Bratislava, Department of Organization and Management of Pharmacy; Martin Hulin, Ing., Mgr., PhD., Study Chair — Research Institute for Child Psychology and Pathopsychology
Locations (24):
- Slovakia (24):
  - Lekáreň Needham, Banská Bystrica
  - Lekáreň V KAUFLANDE BB, s.r.o., Banská Bystrica
  - Lekáreň DANUBIA, Bratislava
  - Lekáreň Dr.Max 12, Bratislava
  - Lekáreň Poliklinika Šustekova, Bratislava
  - Lekáreň GREEN-STRAP, Dubnica nad Váhom
  - Lekáreň Námestie Matice Slovenskej, Dr. Max, Dubnica nad Váhom
  - Lekáreň Dr.Max 90, Nemocnica s poliklinkou Sv.Lukáša, Galanta
  - Lekáreň REDMOON, Hnúšťa
  - Lekáreň 17, Kežmarok
  - Lekáreň Námestie Osloboditeľov, Dr. Max, Liptovský Mikuláš
  - Lekáreň RED-MARKET s.r.o., Malacky
  - Lekáreň PRED NEMOCNICOU, Martin
  - Lekáreň, OC Tulip, Martin
  - Lekáreň Námestie Slobody, Dr. Max, Piešťany
  - Lekáreň HEALTHSTORE, Prešov
  - Lekáreň Dr.Max 22, Rimavská Sobota
  - Lekáreň Dr.Max 36, Rožňava
  - Lekáreň OC Madaras Dr. Max, Spišská Nová Ves
  - Lekáreň EURO FARMÁCIA s.r.o., Trenčín
  - Lekáreň SD5 s.r.o., Trenčín
  - Lekáreň CASTILION, Vranov nad Topľou
  - Železničná Lekáreň, Zvolen
  - Lekáreň Bernolákova, Dr. Max, Žilina

IPD SHARING:
Plan to Share IPD: Yes
All collected data will be anonymized and made available on via Open Science Framework

REFERENCES:
- [Background] Haramiova Z, Stasko M, Hulin M, Tesar T, Kuzelova M, Morisky DM. The effectiveness of daily SMS reminders in pharmaceutical care of older adults on improving patients' adherence to antihypertensive medication (SPPA): study protocol for a randomized controlled trial. Trials. 2017 Jul 18;18(1):334. doi: 10.1186/s13063-017-2063-8. PMID 28720121
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- See also: PRECIS-2 Index — https://www.precis-2.org/Trials/251/Scores